CLINICAL TRIAL: NCT00856362
Title: An Open-label, Single-Dose, 4-Period, Sequential Study to Determine the Effect of Moxidectin on CYP3A4 Activity in Healthy Subjects Using Midazolam as a Probe Substrate
Brief Title: Study Evaluating The Co-Administration Of Moxidectin And Midazolam In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3110A1-1004
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Healthy Subjects
MeSH Terms: interventions — moxidectin; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Moxidectin; Drug: Midazolam

INTERVENTIONS:
Drug: Moxidectin
Drug: Midazolam

SUMMARY:
The purpose of this study is to evaluate the effect of single doses of midazolam on the plasma concentration of a single dose of moxidectin in healthy young adult subjects, and to assess the safety of co-administration of moxidectin and midazolam.

ELIGIBILITY:
Inclusion criteria:

1. Men or women of nonchildbearing potential (WONCBP) aged 18 to 50 years inclusive at screening.

   WONCBP may be included if they are either surgically sterile (hysterectomy and/or oophorectomy) or postmenopausal for ≥1 year (with follicle-stimulating hormone [FSH] ≥38 mIU/mL) and must have a negative pregnancy test result within 48 hours before administration of test article. Women who are surgically sterile must provide documentation of the procedure by an operative report or by ultrasound. Sexually active men must agree to use a medically acceptable form of contraception during the study and continue it for 12 weeks after test article administration.
2. Body mass index in the range of 18 to 30 kg/m2 and body weight ≥50 kg.
3. Healthy as determined by the investigator on the basis of screening evaluations.

Exclusion criteria:

1. Women of childbearing potential.
2. Presence or history of any disorder that may prevent the successful completion of the study.
3. Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Blood samples will be collected for determination of moxidectin and midazolam plasma concentrations | 4 months

SECONDARY OUTCOMES:
Safety based on adverse event monitoring, physical examinations, vital sign measurements, 12-lead electrocardiograms (ECGs) and routine lab tests | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Berlin, Germany